CLINICAL TRIAL: NCT05596383
Title: THE EFFECT OF VITAMIN D SUPPLEMENTATION ON IMPROVING PANCREAS BETA CELL FUNCTION IN TYPE 2 DIABETES MELLITUS: STUDY OF SOD,IL-6,PDX-1 EXPRESSION, and INSULIN RESISTANCE
Brief Title: Effects of Vitamin D Supplementation on SOD,IL-6 and Insulin Resistance in Type 2 Diabetes Mellitus (DM)
Acronym: DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trisakti University (Other)
Responsible Party: Principal Investigator, dr Alvina Alvina,SpPK, clinical pathology specialist, Trisakti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Trisaktipatklin
Record Dates: First submitted 2022-10-17; First posted 2022-10-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-10

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The study was divided into two groups, the intervention group and the control group. The intervention group received vitamin D 5000 IU/day for 6 months and the control group received a placebo (contains microcrystalline, calcium carbonate, sodium starch) for 6 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Vitamin D, dosage form chewable tablet, dosage 5000 IU, frequency every day, duration six months
  Interventions: Dietary Supplement: Vitamin D 5000 IU
- control group (Placebo Comparator): Placebo (microcrystalline,calcium carbonate, sodium starch), dosage form chewable tablet, frequency every day, duration six month
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D 5000 IU — Intervention vitamin D 5000 IU per day, duration six months, dosage form chewable tablet
  Arms: Intervention group
Dietary Supplement: Placebo — Placebo
  Arms: control group

SUMMARY:
The aim of this intervention clinical study are: evaluation the effect of vitamin D supplementation on anti-oxidant status, inflammation, insulin resistance in patients type 2 diabetes mellitus.

The research question is how the effect of vitamin D supplementation for 3 and 6 months on anti-oxidant status, inflammation and insulin resistance in patients type 2 diabetes mellitus.

The main tasks participants will be asked to do:

* interviews, filling the questionnaires, and giving informed consent after receiving an explanation by the researcher about the purpose of the research
* taking blood for screening examination which includes examination of Serum Glutamic Pyruvic Transaminase (SGPT), albumin, creatinine and blood Ca.
* participant who meet the inclusion and exclusion criteria, performed a physical examination (height and weight) and blood collection for examination 25(OH)D.
* Subjects/participant with vitamin D deficiency and insufficiency will be included in randomization, two groups: the group that received vitamin D3 5,000 IU and the group that received a placebo. Vitamin D 5000 IU and placebo taken daily for 6 months.
* Observations for 3 months and 6 months from the first time supplementation was given.

Treatments they'll be given:

* During the study, the subject's clinical condition will be monitored.
* Subject observations are monitored by telephone or google form to subject or their families

DETAILED DESCRIPTION:
Participant register: Patients type 2 DM aged > 18 years who went to the Community Health Centers Mampang were interviewed, filled out questionnaires, and gave informed consent.Interview by interviewers with at least high school education after being given training first by researchers.

The data is entered in a computer excel table by the researcher. Accuracy, completeness of registration data using the screening form.

Data that contains detailed descriptions of each variable used by the registry:

* Gender: differences in the nature, form, and biological function of men and women that determine differences in reproduction, by interview using a questionnaire and identity card.
* Duration DM: time from the first time being diagnosed DM until the start of the study, expressed in months
* Subject's age: calculated from the time the study began with the date of birth listed on the identity card.

Standard Operating Procedures to address registry operations and analysis activities:

* patient recruitment : Patients type 2 DM aged > 18 years who went to the Community Health Centers Mampang were interviewed.
* data collection: using screening form
* data management : using table excel computer
* data analysis : using Statistical Package for the Social Sciences (SPSS) versi 23
* report for adverse event: using form adverse event Sample size assessment : formula for hypothesis testing the mean difference of two groups Plan for missing data : back up data Statistical analysis plan to address the primary and secondary objectives: normality test (kolmogorov Smirnov), test statistic (T independent test or Mann Whitney test, Anova test)

ELIGIBILITY:
Inclusion Criteria:

* male and female, aged > 18 years
* period of DM ≤ 3 years
* using a single anti-diabetic drug (monotherapy)
* HbA1c > 6,5%

Exclusion Criteria:

* receive insulin therapy
* kidney disease, liver disease
* pregnant and lactating women
* allergy history
* hypercalcemia history
* consumption of vitamin D in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
level of Superoxide Dismutase (SOD) | Change from Baseline at 3 and 6 months
  SOD
Interleukin-6 (IL-6) | Change from Baseline at 3 and 6 months
  IL-6 in monocyte: % (method immunoflowcytometry);
pancreatic and duodenal homeobox 1(PDX-1) expression | Change from Baseline at 3 and 6 months
  PDX-1 expression : ct (method polymerase chain reaction /PCR);
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Change from Baseline at 3 and 6 months
  HOMA-IR : formula (fasting insulin (μIU/mL) x fasting blood glucose (mg/dL)/405

SECONDARY OUTCOMES:
vitamin D level | Change from Baseline at 3 and 6 months
  Vitamin D: ng/mL;
(hemoglobin glycate) HbA1C | Change from Baseline at 3 and 6 months
  HbA1c: % ;
fasting blood glucose | Change from Baseline at 3 and 6 months
  Fasting blood glucose: mg/dL ;
fasting insulin | Change from Baseline at 3 and 6 months
  Fasting insulin: μIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Alvina Alvina, Principal Investigator — Universitas Trisakti
Locations (1):
- Community Health Centers Kecamatan Mampang Prapatan, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mansournia MA, Ostadmohammadi V, Doosti-Irani A, Ghayour-Mobarhan M, Ferns G, Akbari H, Ghaderi A, Talari HR, Asemi Z. The Effects of Vitamin D Supplementation on Biomarkers of Inflammation and Oxidative Stress in Diabetic Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Horm Metab Res. 2018 Jun;50(6):429-440. doi: 10.1055/a-0630-1303. Epub 2018 Jun 8. PMID 29883970
- [Result] Yu Y, Tian L, Xiao Y, Huang G, Zhang M. Effect of Vitamin D Supplementation on Some Inflammatory Biomarkers in Type 2 Diabetes Mellitus Subjects: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Ann Nutr Metab. 2018;73(1):62-73. doi: 10.1159/000490358. Epub 2018 Jun 26. PMID 29945132
- [Result] Al-Sofiani ME, Jammah A, Racz M, Khawaja RA, Hasanato R, El-Fawal HA, Mousa SA, Mason DL. Effect of Vitamin D Supplementation on Glucose Control and Inflammatory Response in Type II Diabetes: A Double Blind, Randomized Clinical Trial. Int J Endocrinol Metab. 2015 Jan 10;13(1):e22604. doi: 10.5812/ijem.22604. eCollection 2015 Jan. PMID 25745497